CLINICAL TRIAL: NCT07101640
Title: Pharmacokinetics, Safety and Preliminary Efficacy Study of Montelukast in Critically Ill Infants With Developing Bronchopulmonary Dysplasia
Brief Title: PK, Safety and Preliminary Efficacy Study of Montelukast in Critically Ill Infants With Developing Bronchopulmonary Dysplasia
Acronym: PRISM
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00114044; R01HD113201 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-08-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Bronchopulmonary Dysplasia (BPD); Premature Births; Critical Illness
Keywords: PK; Pharmacokinetics; bronchopulmonary dysplasia; montelukast
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Critical Illness | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Montelukast Sodium (Experimental): Once daily montelukast dosed at 0.75 mg/kg/day, maximum dose 4mg. 4mg of montelukast mixed in 5mlL breast milk/formula for a concentration of 0.8mg/mL.
  Interventions: Drug: montelukast 4 mg granule
- Placebo (Placebo Comparator): Plain breast milk or formula
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: montelukast 4 mg granule — Montelukast sodium (4 mg oral granules) dissolved into 5mL of breast milk/formula yielding a solution concentration of 0.8mg/mL. Dosed once daily by weight, montelukast (0.75 mg/kg/day) or placebo .
  Other Names: montelukast sodium
  Arms: Montelukast Sodium
Drug: Placebo — Plain breast milk or formula
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn how safe montelukast may be in premature infants at significant risk for Bronchopulmonary Dysplasia (BPD) and to determine how much and how quickly montelukast moves from the stomach into the bloodstream, and how quickly it is removed from the bloodstream.

Data supporting the prospect of montelukast benefit involved 6 previous studies involving 206 preterm infants. The dosing ranged from 0.5 to 2.5 mg/kg/day, which aligns with the proposed initial dose of 0.75 mg/kg/day. Though each previous study had a small population, collectively they reveal montelukast as a promising drug in populations of preterm infants developing BPD and for individual preterm infants who are "developing BPD." Thus, researchers expect clinical benefit for preterm infants in this study.

Despite the benefit-to-risk ratio presented by these previous studies, the optimal dose remains to be determined; thus, this study design and PK analysis will start with the lowest dose that is likely to provide direct benefit to participants.

DETAILED DESCRIPTION:
Multi-center, Prospective, Randomized, Double-masked, Placebo-Controlled Trial Participants (n=28) will be enrolled into a randomized, double-blinded, placebo-controlled trial of once daily montelukast (0.75 mg/kg/day) or placebo (1:1 allotment) for 7 days in critically ill premature infants with developing BPD.

The overall aim is to characterize the pharmacokinetics (PK), short- and long-term adverse events (safety), and respiratory support changes (preliminary efficacy) with montelukast following once daily dosing for 7 days.

Primary: Characterize the PK of montelukast in critically ill premature infants with developing bronchopulmonary dysplasia (BPD).

Secondary: Describe the acute safety profile of montelukast and 2-year developmental progress in critically ill premature infants with developing BPD.

Tertiary: Determine preliminary efficacy of montelukast in critically ill premature infants with developing BPD.

Inpatient participation: Will vary based on gestational age and age at randomization; Up to approximately 60 days (7 days of study drug plus 30 days of post-drug safety monitoring or to 36 weeks postmenstrual age, whichever is longer).

Outpatient participation: Medical and neurodevelopmental follow-up assessments at 6, 12, 18 and 24 months old.

ELIGIBILITY:
Inclusion Criteria

1. Documented informed consent from parent or guardian, prior to study activities
2. Receiving mechanical ventilation [high frequency or conventional] and requiring supplemental oxygen (FiO2 ≥ 30%) at time of randomization
3. <28 weeks' gestational age and <1000 g bodyweight at birth
4. 7 to 28 (inclusive) days postnatal age at the time of first study drug dose
5. Able to tolerate 5 mL of enteral volume

Exclusion Criteria

1. Previous enrollment and dosing in the current PRISM study (NICHD-2023-MON01)
2. Previous exposure to montelukast within 7 days prior to randomization
3. Known allergy to montelukast
4. PI deems infant - prior to enrollment - is not expected to survive
5. Has a disease complication that would preclude safe participation of the participant
6. Increased respiratory support due to intercurrent illness (e.g., sepsis, necrotizing enterocolitis, etc.). Infants should be excluded from the study until after resolution of the acute event
7. Congenital lung and diaphragmatic malformations

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Apparent clearance (CL/F) of montelukast | From enrollment to 14 days post first dose.
  The elimination of montelukast divided by the concentration of montelukast.

SECONDARY OUTCOMES:
Volume of distribution | From first dose of study drug though 7 days post last dose.
  The total amount of montelukast in the body to the concentration in the bloodstream.
Half-life | From first dose of study drug though 7 days post last dose.
  The time that it takes for the concentration of montelukast in blood plasma to reach one-half of its steady-state value (the "plasma half-life").
Area Under Curve (AUC) | From first dose of study drug though 7 days post last dose.
  The concentration of montelukast in blood plasma as a function of time.
Maximum Concentration (Cmax) | From first dose of study drug though 7 days post last dose.
  The maximum (or peak) serum concentration that montelukast achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
Death- Safety | From 30 days post treatment or 36 weeks PMA, whichever is longer; through 24 months of follow-up.
  All infants who die at or before 30 days post treatment or 36 weeks PMA, whichever is longer, will be enumerated by treatment group. Researchers will also summarize by treatment group the percent and cumulative incidence of deaths through 24 months of follow-up.
Serious Adverse Events | At or before 30 days post treatment or 36 weeks PMA, whichever is longer.
  Total SAEs by participants. Researchers will determine the incidence (rate per person-time) and prevalence (percent of each treatment group experiencing an SAE) at or before 30 days post treatment or 36 weeks PMA, whichever is longer.
Total Neuropsychiatric Adverse Events (NPAE) | From first dose to 30 days post treatment or 36-weeks PMA, whichever is longer.
  Researchers will collect safety events of special interest: neuropsychiatric events, including irritability, sedation, apnea, convulsion/seizure, sleep disturbance, tremor and neuropsychiatric event (other). 'Other' will be any event not fitting the previous categories but deemed to be neuropsychiatric in nature by the site principal investigator (PI). For total NPAEs, researchers will determine the incidence (rate per person-time) and prevalence (percent of each treatment arm experiencing an NPAE) for each treatment group. For all safety events researchers will calculate the incidence and prevalence for both the treatment period and for the period to 30 days post treatment or 36-weeks PMA, whichever is longer. Site investigators will determine seriousness and severity for all AEs.
Neonatal Infections | From first dose till at or before 30 days post treatment or 36 weeks PMA, whichever is longer.
  Researchers will determine the prevalence (percent of each treatment group experiencing an infectious adverse event) at or before 30 days post treatment or 36 weeks PMA, whichever is longer. Specific infections will include (but not limited to): upper respiratory infections, pharyngitis, sinusitis, and otitis.
Neurodevelopmental outcomes (Bayley-4) | From first dose through 24 months of age.
  The Bayley Scales of Infant and Toddler Development, Fourth Edition, (often referred to as the Bayley-4) will be completed by a site-based specialist at 24 months of age (range 22 to 26 months). The Bayley-4 is a standardized assessment tool designed to evaluate the developmental functioning of infants and toddlers. Composite scores for each domain are standardized, with a mean of 100 and a standard deviation of 15. Composite scores are also converted into percentile ranks, which indicate the child's performance relative to a normative sample. For instance, a percentile rank of 50 means the child is performing at the average level for their age group.
Neurodevelopmental outcomes (Ages and Stages Questionnaires (ASQ)) | 6 months, 12 months, 18 months, and 24 months
  The Ages and Stages Questionnaires (ASQ) is a developmental screening tool designed to assess the developmental progress of children from one month to 5 ½ years of age. For each of the 5 domains assessed by the ASQ, the minimum score is 0 and maximum score is 60. Higher scores mean better outcome.
Neurodevelopmental outcomes (Child Behavior Checklist (CBCL) | 18 months, 24 months
  The Child Behavior Checklist (CBCL) is a widely used tool for assessing behavioral and emotional problems in children as young as infancy and toddlerhood.
Oxygen saturation index (OSI) | From randomization baseline to day 7 of treatment.
  Oxygen saturation index (OSI) is used to assess the severity of respiratory failure. A higher OSI value indicates worse respiratory compromise. The main OSI endpoint will be the change from randomization baseline to day 7 of treatment.

OTHER OUTCOMES:
Delirium Assessment | From Enrollment until at 36 weeks PMA who remain hospitalized.
  The Cornell Assessment of Pediatric Delirium (CAPD) will be completed in infants at 36 weeks PMA who remain hospitalized. This tool involves scoring based on observations over several hours, rather than a single point in time. A score of 9 or higher typically indicates the presence of delirium.
Clinical Bronchopulmonary Dysplasia (BPD) | From first dose through 36 Week PMA.
  Clinical BPD will be determined and graded based on clinical severity, which will be based on respiratory support (supplemental oxygen or positive airway pressure) needed at 36 weeks' PMA. This outcome will be measured on a 4-level ordinal scale (as a-d below) and on a dichotomous scale (moderate-to-severe BPD vs. no BPD/mild BPD).
  1. No BPD - receiving no respiratory support.
  2. Mild (grade 1) BPD - receiving ≤2 L/min nasal cannula.
  3. Moderate (grade 2) BPD - receiving >2 L/min or non-invasive positive airway pressure.
  4. Severe (grade 3) BPD - receiving invasive mechanical ventilation.
Time on supplemental oxygen | From the time of randomization until 30 days post last dose or 36 week PMA, whichever is longer.
  Duration in days that participant requires supplemental oxygen from the time of randomization.
Time on positive pressure ventilation | From the time of randomization until 30 days post last dose or 36 week PMA, whichever is longer.
  Duration in days that participant requires positive airway pressure (any type of mechanical ventilation or continuous positive airway pressure (CPAP) or high-flow nasal cannula >1 L/min flow) from the time of randomization. Researchers will also collect time specifically requiring mechanical ventilation (conventional ventilation or hi-frequency ventilation).
Death- Efficacy | From first dose till at or before 36 weeks PMA
  All infants who died at or before 36 weeks PMA will be included
Death or moderate (grade 2) to severe (grade 3) BPD | From first dose until 24 months of age. (+/- 2 months)
  All infants who die during the course of the study.

IPD SHARING:
Plan to Share IPD: No